CLINICAL TRIAL: NCT02701140
Title: Ticagrelor And PrEconditioning in Patients With coronaRy Artery diSease
Acronym: TAPER-S
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Italo Porto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Italo Porto, MD, PhD, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Not assigned
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Intervention Model Description: PROBE
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: PROBE
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Active Comparator): Ticagrelor will be given in a loading dose of 180 mg followed by a dose of 90 mg twice daily.
  Interventions: Procedure: Coronary stenting; Procedure: intracoronary ECG recording; Procedure: Coronary Flow reserve; Procedure: Index of Microcirculatory Resistance; Procedure: Fractional Flow Reserve
- Clopidogrel (Active Comparator): Clopidogrel will be given in a loading dose of 600 mg followed by a dose of 75 mg once a day.
  Interventions: Procedure: Coronary stenting; Procedure: intracoronary ECG recording; Procedure: Coronary Flow reserve; Procedure: Index of Microcirculatory Resistance; Procedure: Fractional Flow Reserve

INTERVENTIONS:
Procedure: Coronary stenting — Within 1h after the first PCI, patients will be randomized to either ticagrelor or clopidogrel.
Procedure: intracoronary ECG recording — Measurement of ST segment elevation using intracoronary ECG recording
Procedure: Coronary Flow reserve — measured with an intracoronary pressure/temperature sensor-tipped guidewire
  Other Names: CFR
Procedure: Index of Microcirculatory Resistance — measured with an intracoronary pressure/temperature sensor-tipped guidewire
  Other Names: IMR
Procedure: Fractional Flow Reserve — measurement of Fractional Flow Reserve during hyperemic phase.
  Other Names: FFR

SUMMARY:
The aim of this study is to assess the pleiotropic effects of ticagrelor that could represent possible mechanisms for its beneficial effects on cardiovascular mortality. We will test three different hypotheses:

1. Ticagrelor may increase ischemic preconditioning as compared to clopidogrel in patients with stable coronary disease, showing multivessel coronary artery disease and undergoing staged PCI.
2. Ticagrelor may improve microvascular perfusion in the myocardium of patients with multivessel coronary artery disease undergoing staged PCI.
3. Ticagrelor may exert positive effects enhancing the paracrine modulation, migration, homing and survival of hBMDSC, with a potential impact on the microvascular dysfunction and on the protective response to ischemia (cellular preconditioning).

DETAILED DESCRIPTION:
Ticagrelor is a reversibly binding, direct-acting, oral P2Y12 antagonist used for prevention of atherothrombotic events in patients with acute coronary syndrome. It does not belong to thienopyridines; it is a carbocyclic nucleoside, representing a "first-in-class" cyclopentyl-triazolo-pyrimidine.

In 2 phase II studies, dyspnea was noted to occur as a side effect to ticagrelor in a dose-dependent fashion; and in the PLATO study, there was a 6% absolute excess of dyspnea in ticagrelor-treated patients compared with patients treated with clopidogrel. In the ONSET/OFFSET study dyspnea was more commonly associated with ticagrelor therapy in comparison with clopidogrel and placebo in patients with stable coronary artery disease (38.6%, 9.3%, and 8.3%, respectively), but was not associated in this study with any adverse change in cardiac or pulmonary function. This result was confirmed in patients with acute coronary syndrome.

The mechanisms for this side effect are largely unknown, although early data indicate that ticagrelor blocks adenosine reuptake through inhibition of ENT-1 by red blood cells, and it is known that intravenous adenosine infusion can cause transient dyspnea in the absence of bronchoconstriction. Another mechanism potentially increasing adenosine levels by ticagrelor consists in adenosine triphosphate (ATP) release from red blood cells. Moreover, comparison between ticagrelor and adenosine molecules suggests their similarity; Adenosine is a well-known key endogenous molecule that regulates tissue functions by activating 4 G-protein-coupled adenosine receptors: A1, A2A, A2B, and A3. Adenosine accumulates in the extracellular space in response to metabolic stress and cell damage; and elevations of adenosine are found in ischemia, hypoxia, inflammation, and trauma. Adenosine acts as cytoprotector by its anti-inflammatory, cardioprotective, cerebroprotective, antisclerotic, and antifibrotic properties, as well as by platelet inhibition and vasodilation.

It was hypothesized that chronic adenosine overload induced by ticagrelor may contribute to the vascular outcome benefit observed in PLATO, in addition to its inhibitory effect on platelet activity via P2Y12 receptor blockade. Very recently, ticagrelor has been shown to increase adenosine-induced physiological responses in human healthy subjects by shifting the dose-response curve for adenosine-induced coronary blood flow velocity (CBFV) to the left and, in non-ST-segment elevation acute coronary syndrome patients treated with percutaneous coronary intervention and receiving a maintenance dose of ticagrelor, coronary blood flow velocity augments to a greater degree compared with patients on a prasugrel maintenance dose in response to increasing adenosine concentrations. These effects are also compatible with adenosine reuptake blockage, another of the purported pleiotropic effects of ticagrelor. The enhanced ticagrelor-related adenosine bioavailabilty may have beneficial effects through three interrelated mechanisms.

Activation of preconditioning: Ischemic preconditioning, consisting in episodes of ischemia as short as 5 minutes, followed by reperfusion, has been showed to protect the heart from a subsequent longer coronary artery occlusion by markedly reducing the amount of necrosis. Adenosine plays a key role in triggering ischemic preconditioning. Indeed, stimulation of A1 adenosine receptors triggers a complex pathway including the epsilon isoform of protein kinase C, the ATP-dependent potassium channels, the mitochondrial permeability transition pores as well as others, like a paradoxical protective release of oxygen radicals eventually making cells more resistant to ischemia. In humans, examples of preconditioning are the preinfarction angina and the angina "warm-up phenomenon". Preconditioning can be reproduced experimentally by repetitive balloon inflations in the coronary artery that have as principal consequences less chest pain and ST-segment elevation. Pharmacological preconditioning can be induced by intravenous or intracoronary administration of adenosine or A1 agonists of adenosine. In a recent study in rabbits authors observed an anti-infarct effect of clopidogrel and cangrelor (the intravenous analog of ticagrelor) and that it was not the result from blockade of platelet aggregation, but rather from activation of the signal transduction pathway of pre- and postconditioning, involving the reperfusion injury salvage kinases (RISK) including Akt and ERK as well as adenosine A2B receptors, mitochondrial KATP channels, and redox signalingi. This cardioprotective effect of cangrelor was confirmed in a primate model.

Improvement of coronary microvascular dysfunction. Coronary microvascular dysfunction has been demonstrated to affect the prognosis of patients with acute coronary syndromes: Furber et al described that Doppler flow velocity parameters in the infarct-related artery are of prognostic value for long-term cardiac events. Additionally, Takahashi et al. found an impaired coronary flow reserve velocity (CFVR) in the infarct-related artery to be significantly associated with increased cardiac event rates at long-term follow-up. Furthermore, microvascular function has been demonstrated to be altered even in non-ischemic regions at distance from the infarcted myocardial tissue and van de Hoef et al. have recently shown that microvascular dysfunction determined in the reference vessel after percutaneous coronary intervention is associated with a significantly increased long-term cardiac mortality.

Microvascular dysfunction is likely to occur also in the setting of non ST-elevation acute coronary syndromes (NSTEMI): Marzilli et al. found that in patients with unstable angina, episodes of transient myocardial ischemia at rest are associated with a brisk increase in coronary microvascular resistance and that this increase is prevented by the administration of antiplatelet drugs.

Finally, microvascular dysfunction may also occur following successful coronary angioplasty: coronary flow reserve has been shown to be impaired in the vascular bed subtended by the treated artery and requires up to three months for this microvascular dysfunction to resolve.

Activation of cellular preconditioning. Human bone marrow derived stem (hBMDSC) have been shown to have remarkable therapeutic potential in vitro and in vivo. The mechanism of the therapeutic benefits must be multifaceted, involves enhanced expression, and release of trophic/growth factors that provide autocrine and paracrine modulation and protection on the adult human myocardium and stimulation of the endogenous regenerative responses. However, when this class of cells are exposed into an ischemic environment, revealed reduced survival rates and impaired angiogenic capacity. Exposure to sub-lethal hypoxia might impair the intracellular signaling pathways involved in regenerative processes and may not provide a resource of several trophic agents and growth factors that might play important role in cell survival, angiogenesis, and differentiation of hBMDSC. Recently, in animal model of myocardial infarction, P2Y12 blocker cangrelor was shown to be a potent cardioprotective modulator through mobilization of progenitor cells and protective signaling on myocytes and smooth muscle cells rather than any effect on platelet aggregation.

STUDY DESIGN AND METHODOLOGY Hypothesis

The aim of this study is to assess the pleiotropic effects of ticagrelor that could represent possible mechanisms for its beneficial effects on cardiovascular mortality. We will test three different hypotheses:

1. Ticagrelor may increase ischemic preconditioning as compared to clopidogrel in patients with stable coronary disease, showing multivessel coronary artery disease and undergoing staged PCI.
2. Ticagrelor may improve microvascular perfusion in the myocardium of patients with multivessel coronary artery disease undergoing staged PCI.
3. Ticagrelor may exert positive effects enhancing the paracrine modulation, migration, homing and survival of hBMDSC, with a potential impact on the microvascular dysfunction and on the protective response to ischemia (cellular preconditioning).

Study design: The study is a prospective, randomized, open-label, blinded end-point trial that will enroll patients with multivessel, stable coronary artery disease undergoing ischemia-related PCI (evaluated by stress test and/or FFR during coronary catheterization), and requiring staged PCI. Patients that experience an acute coronary syndrome in multivessel coronary artery disease, and that need to complete the revascularization in the non-culprit vessel, may be considered stabilized after one month from the culprit vessel PCI, and therefore may be enrolled. After the procedure the patients should be treated according to local routines. Randomization will be blocked within each study site, in order to get an even balance of patients randomized to either drug within each recruiting center.

The recruitment to the present study will be proposed to 66 consecutive patients and will be submitted for the approval of the local ethics committee and national regulatory authority (AIFA) and will be carried out according to the Italian regulatory rules.

The study will be conducted according to the protocol and in strict compliance with ICH GCP, the Declaration of Helsinki and all applicable regulatory requirements. Before the start of the study, the study protocol, the investigator brochure and other applicable documents will be submitted to independent Ethics Committees (EC) and responsible national and local authorities, as required by each participating country's regulations. The study can start only after the favourable opinion of the EC of the Coordinating Centre. The Coordinating Centre will inform the investigators in writing that all ethical and legal requirements have been met before the first patient is enrolled in the study. After the protocol has been accepted, substantial amendments to this protocol require the approval by the Coordinating Centre. After the end of the study, a final study report will be prepared and distributed to regulatory authorities and ECs as required by applicable regulations. Before a patient can participate in the study, patient's informed consent needs to be obtained according to GCP and the legal requirements of the country concerned. Patient information sheet and consent form must have been reviewed and approved by the responsible EC. The investigator or an authorized designate will explain the nature, purpose, scope and course of the study, including information on the investigational therapy, potential benefits and risks to the patient. In addition to oral information, the patient will receive a written patient information sheet containing all relevant information. Sufficient time will be allowed to discuss any questions raised. Only after this process is completed, consent for participation may be given. Consent must be obtained prior to any study specific procedure and with sufficient time before a study related intervention as per local requirements. The consent form must be personally signed and dated by the individual giving consent and by the investigator or designee who lead the informed consent process with the patient. The consent form must be retained by the investigator as part of the study records. In addition, the patient will receive a copy of the patient information sheet and a copy of his/her signed and dated consent form. Confirmation that consent was obtained will also be documented in the medical records and on the eCRF. Should a protocol amendment be made, the patient information sheet may need to be revised to reflect the change(s) of the protocol. After the EC has approved the revised information sheet and consent form, it is the responsibility of the investigator to inform all active patients affected by the change, and to receive their written consent for continuation in the study.

All patients must be identifiable throughout the study at the study site. The investigator will maintain a personal list of patient numbers and patient names for data reconciliation.

Primary Endpoint: 1) comparison of ticagrelor and clopidogrel on delta (difference) ST-segment elevation by intracoronary ECG during two-step sequential coronary balloon inflation in the culprit vessel;

Secondary Endpoints: 1) comparison of ticagrelor and clopidogrel on CFR, IMR and FFR measured in the culprit vessel and reference vessel at the end of PCI. 2) angina score during coronary balloon inflation.

Statistical analysis and power calculation: Sample size: assuming an absolute difference (delta) of 4 mm in the change of ST-segment shift from the first to the second balloon inflation between the 2 groups, we calculated that 30 patients per group will be required to have an 80% power to detect a statistically significant difference between groups at p < 0.05. Standard deviation (SD) of the primary endpoint is expected to be ~ 5,4 mm in each treatment group. A total of 66 patients will be enrolled considering a total drop-out rate of 10%.

The main analysis to be made is a comparison of the primary and secondary endpoint (continuous variables) between the two groups of 30 patients each, that will be evaluated with Analysis of variance (ANOVA). The co-primary safety endpoint, being a frequency value, will be analysed using Fisher test.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 75 years
* Weight > 60 Kg
* Participants must have read and approved the informed consent and be compliant with the study procedures

Exclusion Criteria:

* Pretreatment (before the first angiogram) with either prasugrel or ticagrelor. Patients initially treated with clopidogrel (including those who had a loading dose) will be enrolled.
* Known hypersensitivity to aspirin, clopidogrel, ticagrelor or any excipients
* Need for concomitant cardiac procedure, such as valve repair or replacement
* Any previous history of ischemic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm)
* Any active pathological bleeding or history of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months, other bleeding diathesis, or considered by investigator to be at high risk for bleeding
* Concomitant oral or IV therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices, (cyclosporine, quinidine), or strong CYP3A inducers (rifampin/rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardia events
* Known pregnancy, breast-feeding, or intend to become pregnant during the study period
* Age < 18 or ≥ 75 years
* Severe uncontrolled chronic obstructive pulmonary disease
* Concomitant theophylline/aminophylline use
* Baseline ECG with infarct or conduction abnormalities (i.e. LVH with repolarization abnormality, bundle branch block, ST-segment abnormalities)
* Evidence of prior myocardial infarction by cardiac imaging
* Depressed left ventricular systolic function at randomization (ejection fraction < 50% within 24 hours after first PCI)
* Clinical congestive heart failure
* Presence of coronary collaterals on diagnostic coronary angiography
* Diffuse obstructive disease (≥ 70% stenosis) in the distal segment of the target vessel
* Left main and/or three-vessel coronary artery disease
* End-stage renal disease
* Known severe hepatic impairment
* Concomitant need for anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
delta (difference) ST-segment elevation by intracoronary ECG | within one hour
  Comparison of ticagrelor and clopidogrel on delta (difference) ST-segment elevation by intracoronary ECG during two-step sequential coronary balloon inflation in the culprit vessel

SECONDARY OUTCOMES:
CFR, IMR and FFR measured in the culprit vessel and reference vessel at the end of PCI | within one hour
  Comparison of ticagrelor and clopidogrel on CFR, IMR and FFR measured in the culprit vessel and reference vessel at the end of PCI
ticagrelor and clopidogrel on angina score | within one hour
  Comparison of ticagrelor and clopidogrel on angina score during coronary balloon inflation.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Amario D, Galli M, Restivo A, Canonico F, Vergallo R, Migliaro S, Trani C, Burzotta F, Aurigemma C, Laborante R, Romagnoli E, Francese F, Ceccarelli I, Borovac JA, Angiolillo DJ, Tavazzi B, Leone AM, Crea F, Patti G, Porto I. Ticagrelor enhances the cardioprotective effects of ischemic preconditioning in stable patients undergoing percutaneous coronary intervention: the TAPER-S randomized study. Eur Heart J Cardiovasc Pharmacother. 2024 May 4;10(3):190-200. doi: 10.1093/ehjcvp/pvad092. PMID 38006237
- [Derived] D'Amario D, Restivo A, Leone AM, Vergallo R, Migliaro S, Canonico F, Galli M, Trani C, Burzotta F, Aurigemma C, Niccoli G, Buffon A, Montone RA, Flex A, Franceschi F, Tinelli G, Limbruno U, Francese F, Ceccarelli I, Borovac JA, Porto I, Crea F. Ticagrelor and preconditioning in patients with stable coronary artery disease (TAPER-S): a randomized pilot clinical trial. Trials. 2020 Feb 17;21(1):192. doi: 10.1186/s13063-020-4116-7. PMID 32066489